CLINICAL TRIAL: NCT07207239
Title: Effect of Theta-burst rTMS Therapy on the Clinical and Cognitive Symptoms of Patients With Therapy Resistant Depression and Response Prediction With Neuroimaging Methods.
Acronym: TMS-DEP-2024
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Gábor Csukly, Associate Professor, Semmelweis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TMS-DEP-2024
Record Dates: First submitted 2025-09-10; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Transcranial Magnetic Stimulation, Repetitive; Depression - Major Depressive Disorder
Keywords: TMS; therapy resistant depression; EEG; MRI; neuroimaging
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TB-rTMS (Experimental)
  Interventions: Device: repetative Transcranial Magnetic Stimulation (rTMS), theta-burst protocol

INTERVENTIONS:
Device: repetative Transcranial Magnetic Stimulation (rTMS), theta-burst protocol — Theta-burst rTMS treatment stimulates the left Dorsolateral Prefrontal Cortex (DLPFC). The TBS parameters the investigators adopted follows the standard TBS protocols, with 3-pulse 50-Hz bursts given every 200 ms (at 5 Hz) and an intensity of 100% active motor threshold. The investigators plan to deliver 1800 stimuli to the left DLPFC daily in 9.5-minute blocks for four weeks.

SUMMARY:
The primary aim of the study is to find the combination of neuroimaging-related markers, demographics, and clinical characteristics that predict the response of patients with therapy-resistant depression to theta-burst rTMS treatment. The secondary aim is to monitor the cognitive effects of TMS therapy.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of depression
2. 18 years of age
3. Beck depression inventory score above 12 (screening)
4. MADRS score above 6 (baseline)

Exclusion Criteria:

1. serious cognitive impairment
2. mental retardation
3. history of head injury with loss of consciousness for more than 1 hour
4. alcohol or drug abuse within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2028-06-13 (Estimated); Study Completion 2028-06-13 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms | 120 days
  The primary outcome measures are the clinical symptoms of depression measured by a clinician with the Montgomery-Åsberg Depression Rating Scale.

SECONDARY OUTCOMES:
Neuroimaging characteristics | 120 days
  A secondary outcome measure is neuroimaging characteristics including the alpha peaks measured by EEG, the nonoscillatory component (1/f) calculated from resting EEG, and connectivity parameters measured by fMRI. These markers will play a part in response prediction.
Patient profile | 120 days
  The patient profile encompasses demographics and clinical characteristics, namely age, sex, level of education, history of other psychiatric conditions, comorbidities, and medications. Together with neuroimaging characteristics, these will be used for response prediction.
Cognitive functioning/Spatial working Memory | 120 days
  The test will be used measure spatial working memory. Memory span is the major outcome variable of this test (the longest number of elements correctly retraced). Higher values indicate better outcomes. Its minimum value is 0 and it has no theoretical maximum value.
Cognitive functioning/Executive function | 120 days
  The test will be used measure executive functioning. Number of mistakes is the major outcome variable of this test (mistakes arise when subjects fail to differentiate a distractor from the continuous task). Higher values indicate worse outcomes. Its minimum value is 0 and it has no theoretical maximum value.
  Time Frame: 120 days
Cognitive functioning/reaction time | 120 days
  The test will be used measure executive functioning and reaction time. Average reaction time is the major outcome variable of this test. Higher values indicate worse outcomes.
Clinical symptoms based on self-report questionnaires | 120 days
  Beck depression inventories are to be used to monitor clinical symptoms of depression

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Budapest, Pest County, Hungary

IPD SHARING:
Plan to Share IPD: No